CLINICAL TRIAL: NCT06801418
Title: A Phase 1, Open-label, Randomized, 2-sequence, 4-period, Fully-replicate, Bioequivalence Study Between Adagrasib Reference Tablets and High Drug Load Tablets in Healthy Adult Participants
Brief Title: Bioequivalence Study Between Adagrasib Reference Tablets and High Drug Load Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0020
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adagrasib sequence A (Experimental)
  Interventions: Drug: Adagrasib
- Adagrasib sequence B (Experimental)
  Interventions: Drug: Adagrasib

INTERVENTIONS:
Drug: Adagrasib — Specified dose on specified days
  Other Names: BMS-986503; MRTX849

SUMMARY:
This is a study to evaluate bioequivalence between adagrasib reference tablets and high drug load tablets in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants without clinically significant deviation from normal in medical history physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory assessments as determined by the investigator.
* Body mass index of 18.0 kg/m2 to 32.0 kg/m^2, inclusive, (BMI may be rounded, eg, a participant with a BMI of 32.4 kg/m^2 would qualify; a participant with a BMI of 32.5 kg/m^2 or higher would not qualify). BMI = weight (kg)/(height [m])^2.
* Total body weight ≥ 50 kg.
* Individuals of childbearing potential (IOCBP) and male (as assigned at birth) participants who are sexually active with IOCBP must agree to follow instructions for method(s) of contraception as included in the ICF.
* A female (as assigned at birth) is eligible to participate if she is not pregnant or breastfeeding and at least 1 of the following conditions applies:

  1. Is not an IOCBP, OR
  2. Is an IOCBP and using a non-hormonal contraceptive method that is highly effective (with a failure rate of < 1% per year).

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, any components of the IMP, or other substance (not including seasonal allergies), unless approved by the investigator and medical monitor.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions.
* History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study, including any of the following:

  i. History of myocardial infarction ii. Heart failure iii. Unstable angina (within 6 months of Day -1) iv. High-risk or symptomatic cardiac arrhythmias (eg, sustained ventricular tachycardia, second- or third-degree atrioventricular block without a pacemaker) v. Hypertension.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve from Time Zero Extrapolated to Infinite Time [AUC(INF)] | Up to Day 28
Area Under the Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)] | Up to Day 28
Maximum Observed Plasma Concentration (Cmax) | Up to Day 28

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) | Up to Day 34
Number of Participants with Clinical Laboratory Test Abnormalities | Up to Day 28
Number of Participants with Vital Sign Abnormalities | Up to Day 28
Number of Participants with Physical Examination Abnormalities | On Day 28
Number of Participants with 12-Lead Electrocardiogram (ECG) Abnormalities | Up to Day 28
Time of Maximum Observed Plasma Concentration (Tmax) | Up to Day 28
Apparent Terminal Phase Half-life (T-HALF) | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 0003, Lenexa, Kansas
  - Local Institution - 0002, San Antonio, Texas
  - Local Institution - 0001, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com